CLINICAL TRIAL: NCT05674747
Title: Pilot Study to Determine the Safety and Efficacy of Regimen Frequencies Using the Swift Microwave Device for Mild to Moderate Toenail Onychomycosis Caused by Dermatophytes
Brief Title: Pilot Study of Swift Microwave Device for Onychomycosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mediprobe Research Inc. (Other)
Collaborators: Emblation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FN1p
Record Dates: First submitted 2022-12-15; First posted 2023-01-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Onychomycosis of Toenail
Keywords: tinea unguium; dermatophyte
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A-Weekly x 4wk (Experimental): Subjects will receive treatment on Day 0 and then weekly in the first month followed by monthly treatment to Month 6 (9 treatments).
  Subjects who do not meet the 'temporary increase in clear nail' criteria at Month 6 and/or Month 9 will be offered once monthly treatment for 3 additional months.
  Interventions: Device: Swift Microwave treatment - weekly x 4wks
- Group B-Biweekly x4wk (Experimental): Subjects will receive treatment on Day 0 and then every two weeks in the first month followed by monthly treatment to Month 6 (7 treatments).
  Subjects who do not meet the 'temporary increase in clear nail' criteria at Month 6 and/or Month 9 will be offered once monthly treatment for 3 additional months.
  Interventions: Device: Swift Microwave treatment - Every other week x 4wks
- Group C-Biweekly x 24wks (Experimental): Subjects will receive treatment on Day 0 and then once every two weeks in the first six months (12 treatments).
  Subjects who do not meet the 'temporary increase in clear nail' criteria at Month 6 and/or Month 9 will be offered once monthly treatment for 3 additional months.
  Interventions: Device: Swift Microwave treatment - Every other week x 24wks

INTERVENTIONS:
Device: Swift Microwave treatment - weekly x 4wks — Swift device set up to 7-9 Watts applied locally for up to a 3 second burst to the toenail.
  Start at 9 Watts and apply locally for up to a 3 second burst; adjust the dose and duration as is tolerable for the subject. Repeat on the infected parts of the nail as is tolerable for the subjects ( up to 5 repetitions).
  Arms: Group A-Weekly x 4wk
Device: Swift Microwave treatment - Every other week x 4wks — Swift device set up to 7-9 Watts applied locally for up to a 3 second burst to the toenail.
  Start at 9 Watts and apply locally for up to a 3 second burst; adjust the dose and duration as is tolerable for the subject. Repeat on the infected parts of the nail as is tolerable for the subjects ( up to 5 repetitions).
  Arms: Group B-Biweekly x4wk
Device: Swift Microwave treatment - Every other week x 24wks — Swift device set up to 7-9 Watts applied locally for up to a 3 second burst to the toenail.
  Start at 9 Watts and apply locally for up to a 3 second burst; adjust the dose and duration as is tolerable for the subject. Repeat on the infected parts of the nail as is tolerable for the subjects ( up to 5 repetitions).
  Arms: Group C-Biweekly x 24wks

SUMMARY:
This is an open, single site, pilot study in Canadian subjects diagnosed with mild to moderate toenail onychomycosis caused by dermatophytes. Three microwave treatment frequencies will be compared for efficacy and safety, evaluated by frequency of treatment-related adverse events, clinical improvement of a treated target toenail and inactivation/elimination of fungus in the target toenail. Outcomes will be evaluated at Month 6, Month 9 and Month 12 after initiation of treatments. Subjects not achieving 'temporary increase in clear nail' at Month 6 may receive extra microwave treatments to Month 9 or Month 12 to improve outcomes.

DETAILED DESCRIPTION:
This is an open, single site, pilot study in Canadian subjects diagnosed with mild to moderate toenail onychomycosis caused by dermatophytes. A total of 45 subjects will be enrolled in the study. All eligible subjects who provide written informed consent will be randomized to one of three groups (15 subjects in each group): Group A, B or C.

The treatment regimen for each group is as follows:

Group A: Subjects will receive treatment on Day 0 and then weekly in the first month followed by monthly treatment for a further 4 months (9 treatments).

Group B: Subjects will receive treatment on Day 0 and then every two weeks in the first month followed by monthly treatment for a further 4months (7 treatments).

Group C: Subjects will receive treatment on Day 0 and then once every two weeks in the first six months (12 treatments).

For all groups, patients not achieving 'FDA efficacy' levels at Month 6 End Visit and/or Month 9 End Visit will be offered continuation of treatments once monthly for 3 months to determine if additional treatment will continue to be safe and increase efficacy. Patients may refuse additional treatment, while continuing in safety follow-up to Months 9/12.

Subjects will be followed up every 3 months for safety and efficacy to Month 12, and at any treatment intervals occurring between these main visits. Efficacy will be assessed by changes in affected nail area and length, both in clinic and through photos. Mycology sampling will be performed at pre-determined intervals to assess fungal presence and viability post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Aged 18 years and above.
3. Not Pregnant or breast feeding.
4. Distal subungual onychomycosis (DSO) in a great toenail.
5. One great toenail as a target for treatment having at least 20% involvement of the nail area and no more than 75% involvement of the nail area.
6. Target toenail thickness 3mm or less.
7. No area of infection < 3mm from the proximal nail fold.
8. Toenail for treatment with fungal infection confirmed by detection of a dermatophyte organism (i.e. Trichophyton rubrum).
9. No more than 4 toenails showing visual signs of onychomycosis, including the target toenail.
10. Subject agrees not to have any oral antifungal treatment or topical onychomycosis treatment during the study.
11. Able to perform study assessments.

Exclusion Criteria:

1. Proximal subungual onychomycosis (PSO).
2. Superficial white onychomycosis (SWO).
3. Nail changes that appear as parallel lines, small pinpoint depressions, brown spots, black or brown linear streaks, complete yellowing of all nails without textural change, green debris below the nail or notches in the nail margin ('non-onychomycotic dystrophy').
4. Nails infected by rare fungal species or non-fungal organisms such as mould or bacteria
5. "Spike" of onychomycosis extending to <3mm from the eponychium (proximal nail fold) of the target toenail.
6. Presence of dermatophytoma (defined as thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail.
7. Patients diagnosed with Diabetes Mellitus (types I and II).
8. Peripheral vascular disease.
9. Recurrent cellulitis.
10. Lymphatic insufficiency.
11. Immunocompromised (due to underlying medical disorders or to immunosuppressive treatments).
12. Exhibit an increased risk of bacterial infections due to skin breakdown induced by a fungus
13. Have a current infection or condition of the feet (fungal or otherwise) which may require antifungal or antibacterial treatment during therapy that may confound the study data.
14. Nails for treatment involving the lunula.
15. Co-morbidities including psoriasis, lichen planus or other medical conditions known to induce nail changes.
16. Patients with trauma from ill-fitting shoes, running or overly-aggressive nail care.
17. Subjects that have podiatric/ nursing nail care on a regular basis.
18. Previous target toenail surgery with any residual disfigurement.
19. Nails infected with Candida.
20. Any uncontrolled condition which, in the opinion of the Investigator, may put the subjects at undue risk of adverse effects during the study.
21. Subjects who have had any topical onychomycosis medication for at least 3-months prior to start of treatment or oral antifungal medication at least 6-months prior to study treatment.
22. Implantable Cardioverter Defibrillator (ICD), pacemaker or other implantable device.
23. Metal implants at the site of treatment (within foot or ankle).
24. Severe moccasin tinea pedis.
25. Known allergy or intolerance to microwave therapy.
26. Subject who has had any topical metallic or ionic treatment (e.g, aluminum chloride, silver nitrate) in the target or treated toenail areas within the last 6 months and agrees not to use any during the study.
27. Current participation in a non-observational trial, or have done so within the last 30-days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Number of patients able to complete treatment regimen per protocol | Month 6
  Proportion of Patients able to complete therapy as planned, and summary list of treatment-related Adverse Events reported cross-referenced to severity (mild/moderate/severe) and resolution frequency (resolved before further treatment with no sequelae).
Proportion of Patients per group with 'Temporary Increase in Clear Nail' | Month 6
  'FDA Efficacy' - regimen meets the FDA definition of 'temporary increase in clear nail' in the Target Toenail:
  1. Evidence of nail improvements noted at End of Month 3 using either clear nail increase measured from proximal nail fold, or by increase in clear nail area,
     AND efficacy at End of Month 6 defined by at least one of the following:
  2. At least 6mm increase in clear nail measured from the proximal nail fold
  3. An additional 60mm2 of clear nail with evidence of outward growth
  4. Complete clearance if less than 6mm distal nail was involved prior to treatment

SECONDARY OUTCOMES:
Number of patients able to complete Long-term treatment | Month 12
  Proportion of Patients able to complete therapy beyond Month 6, if required, and summary list of treatment-related Adverse Events reported cross-referenced to severity (mild/moderate/severe) and resolution frequency (resolved before further treatment with no sequelae).
Proportion of patients achieving End of Month 6 Efficacy | Month 6
  At least one of the following in the Target Toenail:
  1. At least 3mm increase in clear nail measured from the proximal nail fold
  2. A 30% increase in area of clear nail, with evidence of outward growth
Proportion of patients per group with Mycological Cure | Month 6, Month 9, Month 12
  Microscopy negative and culture negative
Proportion of patients per group with Effective Cure | Month 6, Month 9, Month 12
  <=10% affected area in target toenail with mycological cure

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Gupta, MD,PhD, Principal Investigator — Mediprobe Research Inc.
Locations (1):
- Mediprobe Research Inc, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta AK, Cooper EA, Wang T. Safety and efficacy of the swift microwave device in patients with mild-to-moderate onychomycosis: Protocol of an open-label, randomized, dose-finding pilot study. Skin Health Dis. 2024 Oct 10;4(6):e455. doi: 10.1002/ski2.455. eCollection 2024 Dec. PMID 39624747